CLINICAL TRIAL: NCT00343356
Title: Clinical Study of Intravesical Epirubicin Plus BCG to Prevent the Recurrence of Transitional Cell Carcinoma of Bladder After Surgical Management
Brief Title: Intravesical Epirubicin Plus BCG to Prevent the Recurrence of Transitional Cell Carcinoma of Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LanZhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LanZhou University; 1996L01936
Record Dates: First submitted 2006-06-19; First posted 2006-06-22 (Estimated); Last update posted 2006-06-22 (Estimated); Status verified 1996-05

CONDITIONS: Bladder Neoplasms
Keywords: Bladder neoplasm;; Carcinoma;; Epirubicin;; BCG;; Perfusion
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma

INTERVENTIONS:
Drug: Trement

SUMMARY:
Biochemotherapy (combined immunotherapeutic drugs and chemotherapeutic drugs) has shown virtue than that use chemical or biological drugs alone in the treatment of some malignant tumor. Here we investigated the efficacy of sequential intravesical therapy with EPI and BCG to EPI or BCG alone in patients with transitional cell carcinoma of bladder cancer after surgical management.

DETAILED DESCRIPTION:
Methods From July 1996 to November 2003, a total of 138 cases of bladder cancer underwent TURBT or partial cystectomy were entered the trail. They were divided into 3 groups randomly: 1, EPI plus BCG; 2, use BCG alone; and 3, use EPI alone. All the patients have been followed up for 28-40 months after surgery (average time was 36 months), and the frequency of bacterial, chemical cystitis and other local side effects were also observed.Results After a median follow up of 36 months, the number of recurrences in group 1 was significantly reduced than group 2 and 3 (p<0.05 vs group 2 and 3, x2-test). The frequency of bacterial, chemical cystitis and other local side effects was similar in group 1 and 2, whereas significant severe side effect was found in group 3 (p<0.05 vs group 2 and 1, x2-test). Allergic reactions, including skin rash, were more frequent in group 3, and other systemic effects were more frequent in group 1. Conclusion Biochemotherapy by single dose EPI plus sequential BCG intravesical is markedly effect in preventing the recurrence of bladder cancer after surgical management. Its side effects are low. This method is of high clinical value.

ELIGIBILITY:
Inclusion Criteria:

* primary single or multiple (more than 2 tumors) pTa to pT1 transitional cell carcinoma, solitary or multiple grade Ⅲ tumors and primary or concomitant carcinoma in situ of the bladder were included in the study

Exclusion Criteria:

* Previous radiotherapy, intravesicial or systemic chemotherapy within 3 months of the study, presence of a second primary malignancy and transitional cell carcinoma of the upper urinary tract or prostatic urethra, invasion of periurethral prostatic ducts, prostatic gland or stroma were exclusion criteria

Ages: 26 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 1996-06; Study Completion 2003-07

PRIMARY OUTCOMES:
Recurrence rate

SECONDARY OUTCOMES:
Side effect: Local toxicity was defined as the occurrence of culture proved bacterial cystitis, chemical or drug-induced cystitis, or other local side effects, such as hematuria, prostatitis or epididymiti

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xiangbo, Principal Investigator — Lanzhou University Second Hospital

REFERENCES:
- [Background] Calais da Silva F, Denis L, Bono A, Bollack C, Bouffioux C. Intravesical chemoresection with 4'-epi-doxorubicin in patients with superficial bladder tumors. Eur Urol. 1988;14(3):207-9. doi: 10.1159/000472938. PMID 3289935
- [Background] Rintala E, Jauhiainen K, Rajala P, Ruutu M, Kaasinen E, Alfthan O. Alternating mitomycin C and bacillus Calmette-Guerin instillation therapy for carcinoma in situ of the bladder. The Finnbladder Group. J Urol. 1995 Dec;154(6):2050-3. PMID 7500456